CLINICAL TRIAL: NCT02380625
Title: An Adaptive Randomized Trial Comparing Multiple Treatments for Ebola Virus (EBOV) Infected Children and Adults
Brief Title: Multiple Treatments for Ebola Virus Disease (EVD)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Clinical Research Management, Inc. (Industry)
Collaborators: Bill and Melinda Gates Foundation (Other); Duke University (Other); University of Sierra Leone (Other); Syneos Health (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVD-003
Record Dates: First submitted 2015-03-01; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Ebola Virus Disease
Keywords: Ebola; EVD; Adaptive design; therapeutics
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Azithromycin; Sunitinib; Erlotinib Hydrochloride; Atorvastatin; Irbesartan; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Azithromycin (Experimental): Azithromycin, IV fluids and laboratory testing
  Interventions: Drug: Azithromycin; Other: IV fluids and laboratory testing
- Sunitinib and Erlotinib (Experimental): Sunitinib, Erlotinib, IV fluids and laboratory testing
  Interventions: Drug: Sunitinib and Erlotinib; Other: IV fluids and laboratory testing
- Atorvastatin and Irbesartan (Experimental): Atorvastatin, Irbesartan, IV fluids and laboratory testing
  Interventions: Drug: Atorvastatin and Irbesartan; Other: IV fluids and laboratory testing
- IV fluids and laboratory testing (Other): no additional treatment
  Interventions: Other: IV fluids and laboratory testing

INTERVENTIONS:
Drug: Azithromycin — Adults (>18 yrs): 3 x 500mg tablets daily for 5 days; Children (6 months to <18 yrs): 30mg/kg (oral suspension) daily for 5 days
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Sunitinib and Erlotinib — Sunitinib - Adults (>18 yrs): 1 x 50mg tablet daily for 7 days; Children (6 months to <18 yrs): 0.83 mg/kg (oral suspension) daily for 7 days. Erlotinib - Adults (>18 yrs): 1 x 150mg tablet daily for 7 days; Children (8kg to <20kg): 3.5 mg/kg daily for 7 days; Children (>20kg to <30kg): 3.0 mg/kg daily for 7 days; Children (>30kg to < 18 yrs): 25 mg/kg daily for 7 days
  Other Names: Sutent; Tarceva
  Arms: Sunitinib and Erlotinib
Drug: Atorvastatin and Irbesartan — Atorvastatin - Adults (>18 yrs): 1 x 40mg tablet daily until discharge; Children (6 years to <18 yrs): 1 x 40mg tablet daily until discharge; Irbesartan - Adults (>18 yrs): 1 x 150mg tablets daily until discharge; Children (6 years to <18 yrs): 1 x 75mg tablet daily until discharge.
  Other Names: Lipitor; Avapro
  Arms: Atorvastatin and Irbesartan
Other: IV fluids and laboratory testing — All arms will receive aggressive IV fluid rehydration and frequent laboratory tests to assist with medical management as indicated.

SUMMARY:
The purpose of this study is to determine whether multiple therapeutic regimens are effective in the treatment of Ebola Virus Disease (EVD)

DETAILED DESCRIPTION:
The ongoing epidemic of EVD has ravaged parts of West Africa, with initial cases reported in December 2013. There is no licensed specific therapy for the disease, which has a case-fatality rate of approximately 50-70%. Although anecdotal clinical data, recent studies in animal models, and in vitro screening suggest that treatment of EVD patients with anti-viral agents, immune modifying agents, and/or convalescent blood products may be effective, they have not been evaluated in clinical trials. This multi-arm clinical trial will evaluate the efficacy and safety of multiple regimens, both as mono-therapy and combination therapy. Provision of these regimens, if found effective and safe, would have a major impact on the current and future epidemics by providing effective treatment options.

As described for previous adaptive trials, a randomization probability for each of the treatment regimens is created based on 14-day mortality, and is used for weighting randomization of subsequently enrolled participants. Participants will continually be preferentially assigned to regimens with better initial performance. New agents can be added or existing agents removed as the trial evolves.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 6 months and >8kg in weight
* Confirmed case of EVD
* Admission to the hospital < 48 hours prior to enrollment
* Participant or family member/guardian able and willing to provide signed informed consent

Exclusion Criteria:

* Prior treatment with any other specific experimental anti-EVD product, or expectation to receive another experimental anti-EVD product during the course of the study (this does not include general supportive care or nutritional supplements routinely administered to all hospitalized patients with EVD)
* Unresponsive
* In the treating physicians opinion, an inability to comply with the study treatment regimen

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Death by 14 days | 14 days after starting treatment regimen

SECONDARY OUTCOMES:
Reduction in viral load | 14 days after starting treatment regimen
2-week post discharge clinical sequelae, including signs and symptoms and laboratory abnormalities | 14 days after starting treatment

OTHER OUTCOMES:
Severe adverse events that are inconsistent with EVD and are assessed as related to study agent(s) by the site principal investigator | 14 days after starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Woods, MD, MPH, Principal Investigator — Duke University; John M Griffiss, MD, Study Chair — Clinical Research Management; David L Hoover, MD, Study Chair — Clinical Research Management

REFERENCES:
- [Derived] Berry SM, Petzold EA, Dull P, Thielman NM, Cunningham CK, Corey GR, McClain MT, Hoover DL, Russell J, Griffiss JM, Woods CW. A response adaptive randomization platform trial for efficient evaluation of Ebola virus treatments: A model for pandemic response. Clin Trials. 2016 Feb;13(1):22-30. doi: 10.1177/1740774515621721. Epub 2016 Jan 14. PMID 26768569